CLINICAL TRIAL: NCT05011422
Title: A Pilot Study of Haploidentical Hematopoietic Stem Cell Transplantation With Ex Vivo TCR Alpha/Beta and CD19 Depletion in Pediatric Hematologic Malignancies
Brief Title: Haploidentical Hematopoietic Stem Cell Transplantation With Ex Vivo TCR Alpha/Beta and CD19 Depletion in Pediatric Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202203051
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Hematologic Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Recipients: ex vivo αβ-TCR/CD19 depleted haplo-hematopoietic stem cell infusion (HSCT) (Experimental): * Patients will undergo standard of care conditioning regiment prior to HSCT
  * On Day 0, patients will undergo infusion of the ex vivo αβ-TCR/CD19 depleted haplo-HSCT from a stimulated peripheral stem cell source per institutional standard of care. Patients whose graft has a residual CD20+ count > 1.0 x 10^5 may receive a single infusion of rituximab on Day +1 at a dose of 375 mg/m^2 at provider's discretion.
  Interventions: Device: Ex Vivo T-cell receptor alpha-beta and CD19+ Depletion using CliniMACs Plus
- Donors: (No Intervention): Donors who meet the eligibility criteria will be mobilized as per institutional standard practice using G-CSF 10 mcg/kg/day with leukapheresis to take place on Day 5. The target volume for collection is 20 L. Up to 4 days of pheresis are permitted to ensure target collection.

INTERVENTIONS:
Device: Ex Vivo T-cell receptor alpha-beta and CD19+ Depletion using CliniMACs Plus — Once pheresed, the product will be washed to remove platelets and the cell concentration will be adjusted per laboratory and ClinicMACS technology recommendations. It is then labeled using the CliniMACS αβ-TCR Biotin Kit and CD19+ immunomagnetic microbeads. After labeling, the cells are washed to remove unbound microbeads. The partially processed product is loaded on the CliniMACS device where labeled cells are depleted and the negative fraction is eluted off the device. The negative fraction is centrifuged and volume reconstituted to obtain the final product
  Arms: Recipients: ex vivo αβ-TCR/CD19 depleted haplo-hematopoietic stem cell infusion (HSCT)

SUMMARY:
This single arm pilot phase I study with safety run-in is designed to estimate the safety and efficacy of a familial mismatched or haploidentical hematopoietic stem cell transplantation (haplo-HSCT) using a novel graft modification technique (selective αβ-TCR and CD19 depletion).

ELIGIBILITY:
Recipient Inclusion Criteria:

* Must meet at least one of the following disease criteria:

  * B cell ALL in first remission and any of the following:

    * Persistent flow-based MRD at end-of-consolidation:

      * ≥ 1% for NCI SR ALL
      * ≥ 0.01% for NCI HR ALL
    * TCF3-HLF t(17;19)
    * KMT2A rearranged infant ALL, < 6 months of age and presenting WBC of > 300,000 or poor steroid response (peripheral blasts >= 1000 /uL on day 8 of therapy
    * Other high-risk features not explicitly stated here, after discussion/approval with protocol PI.
  * B cell ALL in second remission and any of the following:

    * Early (<36 months from start of therapy) marrow or combined relapse
    * Late (>36 months from start of therapy) marrow or combined relapse with end-of re-induction flow MRD >= 0.1%
    * Early isolated extramedullary relapse (< 18 months from start of therapy)
  * Any B cell ALL in third or greater remission
  * T cell ALL in first remission

    * End-of consolidation MRD > 0.1%
  * Any T cell ALL in second or greater remission
  * AML in first remission with any of the following high-risk features:

    * MRD ≥ 1% after first induction course
    * MRD ≥ 0.1% after second induction course
    * RPN1-MECOM
    * RUNX1-MECOM
    * NPM1-MLF1
    * DEK-NUP214
    * KAT6A-CREBBP (if >= 90 days at diagnosis)
    * FUS-ERG
    * KMT2A-AFF1
    * KMT2A-AFDN
    * KMT2A-ABI1
    * KMT2A-MLLT1
    * 11p15 rearrangement (NUP98 - any partner gene)
    * 12p13.2 rearrangement (ETV6 - any partner gene)
    * Deletion 12p to include 12p13.2 (loss of ETV6)
    * Monosomy 5/Del(5q) to include 5q31 (loss of EGR1)
    * Monosomy 7
    * 10p12.3 rearrangement (MLLT10b - any partner gene)
    * FLT3/ITD with allelic ratio > 0.1%
    * RAM phenotype as evidenced by flow cytometry: bright CD56+, dim to negative CD45 and CD38 and lack of HLA-DR
    * Other high-risk features not explicitly stated here, after discussion/approval with protocol PI.
  * AML in second or greater remission
  * Mixed phenotype or undifferentiated leukemia in any CR
  * Secondary to therapy-associated leukemia in any CR
  * NK cell lineage leukemia in any CR
  * Myelodysplastic syndrome (MDS)
  * Juvenile myelomonocytic leukemia (JMML)
* May have undergone a prior hematopoietic stem cell transplant provided one of the criteria in Inclusion Criterion #1 are met AND the patient does not have active GVHD (has been off immunosuppression for at least 3 months).
* Available familial haploidentical donor.
* Donor and recipient must be identical at a minimum of one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. A minimum of 5/10 match is required and will be considered sufficient evidence that the donor and recipient share one HLA haplotype.
* No more than 30 years of age
* Lansky or Karnofsky performance status > 50%
* Adequate organ function as defined below:

  * Cardiac: LVEF ≥ 40% at rest or SF ≥ 26%
  * Hepatic:

    * Total bilirubin < 3 x IULN for age
    * AST(SGOT)/ALT(SGPT) < 5 x IULN
  * Renal: GFR ≥ 60 mL/min/1.73m2 as estimated by updated Schwartz formula for ages 1-17 years (see Appendix B), 24-hour creatinine clearance, or renal scintigraphy. If GFR is abnormal for age based on updated Schwartz formula, accurate measurement should be obtained by either 24-hour creatinine clearance or renal scintigraphy. Renal function may also be estimated by serum creatinine based on age/gender. A minimum serum creatinine of 2x upper limit of normal is required for inclusion on this protocol.
  * Pulmonary:

    * O2 saturation ≥ 92% on room air without positive pressure support
    * FEV1, FVC, and DLCO ≥ 50% of predicted (for children unable to perform a pulmonary function test, a high-resolution CT chest may be obtained)
* The effects of these treatments on the developing human fetus are unknown. For this reason, patients of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for 24 months following transplant. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Recipient Exclusion Criteria:

* Available matched related donor. A patient with a matched unrelated donor is eligible if urgent transplantation is required. A prior unrelated donor search is not required for enrollment.
* Active non-hematologic malignancy. History of other malignancy is acceptable as long as therapy has been complete and there is no evidence of disease.
* Currently receiving any other investigational agents at the time of transplant.
* Active CNS or extramedullary disease. History of CNS or extramedullary disease now in remission is acceptable.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to conditioning agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (bacterial, viral with clinical instability, or fungal), symptomatic congestive heart failure, or unstable cardiac arrhythmia.
* Presence of significant anti-donor HLA antibodies per institutional standards. Anti-donor HLA Antibody Testing is defined as a positive crossmatch test of any titer (by complement dependent cytotoxicity or flow cytometric testing) or the mean fluorescence intensity (MFI) of any anti-donor HLA antibody by solid phase immunoassay.
* Presence of a second major disorder deemed a contraindication for HSCT.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of the start of conditioning.

Donor Eligibility Criteria:

* At least 6 months of age
* Meets the selection criteria as defined by the Foundation for the Accreditation of Hematopoietic Cell Therapy (FACT).
* Able to understand and willing to sign an IRB-approved written informed consent document (or that of legally authorized representative, if applicable).

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the number of events occurring within the first 100 days post-transplant | Through 100 days post-transplant
  -Events are death, disease recurrence or progression, and graft failure
Engraftment as measured by time to neutrophil count recovery | From day of transplant (day 0) to 42 days (+/- 14 days) post transplant
  Time to neutrophil recovery is defined as the first of 3 measurements on different days when the patient has an absolute neutrophil count of >500/μL after conditioning.
Engraftment as measured by time to platelet count recovery | From day of transplant (day 0) to 75 days (+/- 14 days) post transplant)
  Time to platelet recovery is defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count > 50,000/μL AND did not receive a platelet transfusion in the previous 7 days. The exception is the case in which a patient receives platelet transfusions specifically to achieve a higher platelet threshold to allow for an invasive procedure or protection if determined to be at elevated bleeding risk.
Donor cell chimerism as measured by short tandem repeat analysis | Through day +100
  * Can use peripheral blood samples or bone marrow samples
  * The percent of donor-derived cells are sequentially followed.

SECONDARY OUTCOMES:
Event free survival (EFS) | At 24 months post transplant
  -Death, disease recurrence or progression, and graft failure are considered events
Overall survival (OS) | At 24 months post transplant
  Death by any cause is considered an event.
Incidence of grade IV acute GVHD | Weekly through day +100
  -Graded according to the NIH consensus criteria.
Incidence of severe chronic GVHD | Day 101 through 24 months
  -Graded according to the NIH consensus criteria.
Change in Lansky/Karnofsky performance score | Day +100, Day +180, Day +365, and +24 months
  * Lansky is used for participants <15.99 years of age
  * Karnofsky is used for participants >16.00 years of age
Number of pulmonary toxicities | Through 24 months
Number of neurologic/neurocognitive toxicities | Through 24 months
Number of cardiac toxicities | Through 24 months
Number of renal toxicities | Through 24 months
Number of hepatic toxicities | Through 24 months
Number of metabolic toxicities | Through 24 months
Number of thyroid toxicities | Through 24 months
Incidence and severity of acute GVHD | From day +14 through Day +100
  -Graded according to the NIH consensus criteria.
Incidence and severity of chronic GVHD | From day +101 through 24 months
  -Graded according to the NIH consensus criteria.
Number of participants with infections requiring hospitalizations | Through 24 months
Immune reconstitution as measured by recovery of absolute neutrophil count | Over 24 months
Immune reconstitution as measured by recovery of absolute monocyte count | Over 24 months
Immune reconstitution as measured by regain of function of NK cell populations | Over 24 months
  * Immune reconstitution is defined as regain of function of donor-derived immunogenic cells. Immune reconstitution is to be measured by recovery of individual cellular compartments
  * Via flow cytometry
Immune reconstitution as measured by regain of function of T cell populations | Through 24 months
  * Immune reconstitution is defined as regain of function of donor-derived immunogenic cells. Immune reconstitution is to be measured by recovery of individual cellular compartments
  * Via flow cytometry
Immune reconstitution as measured by regain of function of B cell populations | Through 24 months
  * Immune reconstitution is defined as regain of function of donor-derived immunogenic cells. Immune reconstitution is to be measured by recovery of individual cellular compartments
  * Via flow cytometry
Immune reconstitution as measured by regain of function of immunoglobulin G (IgG) | Over 24 months
  * Immune reconstitution is defined as regain of function of donor-derived immunogenic cells. Immune reconstitution is to be measured by recovery of individual cellular compartments
  * Via serum analysis
Immune reconstitution as measured by regain of function of immunoglobulin A (IgA) | Over 24 months
  * Immune reconstitution is defined as regain of function of donor-derived immunogenic cells. Immune reconstitution is to be measured by recovery of individual cellular compartments
  * Via serum analysis
Immune reconstitution as measured by regain of function of immunoglobulin M (IgM) | Over 24 months
  * Immune reconstitution is defined as regain of function of donor-derived immunogenic cells. Immune reconstitution is to be measured by recovery of individual cellular compartments
  * Via serum analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bednarski, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu